CLINICAL TRIAL: NCT00239317
Title: Tamsulosin Phase III Clinical Trial -Double-Blind, Placebo Controlled Study in Male Patients With Lower Urinary Tract Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B617/LCT3
Record Dates: First submitted 2005-09-19; First posted 2005-10-17 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Urinary Tract Diseases
Keywords: tamsulosin; urinary tract diseases; male
MeSH Terms: conditions — Urologic Diseases

INTERVENTIONS:
Drug: Tamusulosin

SUMMARY:
The purpose of this study is to determine whether Tamusulosin is effective in the treatment of lower urinary tract syndrome with male patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urination disorder not accompanied by apparent organic or neurologic abnormality(lower urinary tract syndrome: LUTs).

Exclusion Criteria:

* Patients with urination disorder accompanied by apparent organic(benign prostatic hyperplasia: BPH) or neurologic abnormality, active urinary tract infections, severe cardiovascular, hepatic and/or kidney complications.

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Clinical Development, Astellas Pharma Inc.
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Touhoku Region